CLINICAL TRIAL: NCT06636396
Title: Feasibility of Measuring Skin Carotenoid Level in an Asthma Clinic
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dave Burnett, Associate Professor, University of Kansas Medical Center
Other Study IDs: STUDY00147843
Record Dates: First submitted 2021-11-12; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to assess the use of a practical tool to objectively measure the fruit and vegetable intake in people with asthma.

DETAILED DESCRIPTION:
After consenting to join the study, all participants enter a single cohort, cross-sectional study to assess pulmonary function, asthma control, carotenoid level, and diet intake.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary patients 18 years of age and older
* Confirmed diagnosis of asthma by a physician and confirmed by a pulmonary physician
* English speaking
* Access to the internet

Exclusion Criteria:

* Acute upper or lower respiratory infection
* Systemic corticosteroids
* Recent or current confirmed diagnosis of Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All people with asthma who are at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
FEV1 | measured at a single time point when recruited in the study (cross sectional). Study outcomes will be reported upon study completion, approximately 1 year from study onset.
  forced expiratory volume in one second
ACT | measured at a single time point when recruited in the study (cross sectional). Study outcomes will be reported upon study completion, approximately 1 year from study onset.
  Asthma control test results in a score of 5-25, with a lower score indicating better asthma control.
Skin Carotenoid Level | measured at a single time point when recruited in the study (cross sectional). Study outcomes will be reported upon study completion, approximately 1 year from study onset.
  Skin carotenoid level, measured with a non-invasive tool and is an indicator of fruit and vegetable intake. Skin carotenoid levels are shown as a score of 0-800, with a higher score representing a higher level of carotenoids.
Diet Intake | measured at a single time point when recruited in the study (cross sectional). Study outcomes will be reported upon study completion, approximately 1 year from study onset.
  Nutrascreen diet questionnaire to assess nutritional intake. Specifically, quantity of fruits and vegetable intake will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Burnett, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No